CLINICAL TRIAL: NCT01782976
Title: A Phase II Trial of Cilengitide Plus Bevacizumab in Patients With Recurrent Glioblastoma
Brief Title: Ph II Cilengitide Plus Bevacizumab for Recurrent Glioblastoma (GBM)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Brain Tumor Trials Collaborative (Other); EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTTC11-04
Record Dates: First submitted 2013-01-31; First posted 2013-02-04 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GBM; Intracranial glioblastoma; Recurrent; MD Anderson Symptom Inventory for Brain Tumors; MDASI-BT; Questionnaire; Survey
MeSH Terms: conditions — Glioblastoma; Recurrence | interventions — Cilengitide; Bevacizumab; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cilengitide + Bevacizumab (Experimental): Cilengitide administered intravenously at 2000 mg twice weekly, while Bevacizumab administered intravenously at 10 mg/kg every other week. Each cycle of therapy will be 4 weeks long.
  Interventions: Drug: Cilengitide; Drug: Bevacizumab; Behavioral: Questionnaire

INTERVENTIONS:
Drug: Cilengitide — 2000 mg by vein twice weekly of each 28 day cycle.
  Other Names: EMD 121974
Drug: Bevacizumab — 10 mg/kg by vein on Days 1 and 15 of each 28 day cycle.
  Other Names: Avastin; Anti-VEGF monoclonal antibody; rhuMAb-VEGF
Behavioral: Questionnaire — Completion of MD Anderson Symptom Inventory for Brain Tumors (MDASI-BT) at baseline, Day 1 of cycle 2, and at end of treatment visit. Questionnaire should take about 5 minutes to complete.
  Other Names: Survey

SUMMARY:
The goal of this clinical research study is to learn if cilengitide given in combination with bevacizumab can help to control glioblastoma. The safety of this drug combination will also be studied.

Cilengitide is designed to block the flow of blood to cancer cells, which may help to slow or block the growth of cancer.

Bevacizumab is designed to block the growth of new blood vessels, which may help to slow or block the growth of cancer.

DETAILED DESCRIPTION:
Study Drug Administration:

Each study cycle is 4 weeks. The length of any study cycle may be extended if you experience side effects from the drugs.

Cilengitide will be given as an intravenous (IV) infusion (into a vein) 2 times a week during each 4-week cycle. The infusion will last about 1 hour each time and will be separated by at least 72 hours.

Bevacizumab will be given on as an IV infusion over 90 minutes on Days 1 and 15 of each cycle. After several infusions and depending on how you react, the length of time of the infusion may decrease.

If the study doctor thinks it is in your best interest and depending on how you react to bevacizumab, the length of the infusion time may be decreased.

On the days you are scheduled to receive both cilengitide and bevacizumab, you will receive cilengitide after the bevacizumab infusion.

Study Visits:

On Day 1 of Cycle 1, urine and blood (about 1 tablespoon) will be collected for routine tests.

On Day 15 of Cycle 1, your blood pressure will be measured and blood (about 1 tablespoon) will be drawn for routine tests.

Day 1 of Cycles 2 and beyond:

* You will have a physical exam including measurement of your weight and vital signs.
* Your performance status will be recorded.
* You will complete the MDASI-BT questionnaire.
* Urine and blood (about 1 tablespoon) will be drawn for routine tests.
* You will have a CT or MRI scan to check the status of the disease (only at Cycles 2, 4, 6, 8, and so on.)

On Day 15 of Cycles 2 and beyond, your blood pressure will be measured.

End-of-Treatment Visit:

After your last dose of the study drugs, you will have and end-of-treatment visit and the following tests and procedures will be performed:

* You will have a physical exam including measurement of your weight and vitals.
* Your performance status will be recorded.
* You will have a neurologic exam.
* Your performance status will be recorded.
* You will complete the MDASI-BT questionnaire.
* Urine and blood (about 1 tablespoon) will be collected for routine tests.
* You will have a CT or MRI scan to check the status of the disease.

Length of Treatment:

You may continue taking the study drugs for as long as the doctor thinks it is in your best interest. You will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the long-term follow-up phone calls.

Long-Term Follow-Up Visit:

After you have stopped taking the study drugs and completed your end-of-treatment visit, the study staff will call you 1 time every 6 months to check on how you are doing. Each phone call should last about 5 minutes.

This is an investigational study. Bevacizumab is FDA approved and commercially available for the treatment of recurrent glioblastoma. Cilengitide is not FDA approved or commercially available. At this time, the combination of cilengitide and bevacizumab is being used for research purposes only.

Up to 39 participants will take part in this multicenter study. Up to 20 will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven intracranial glioblastoma (GBM) will be eligible for this protocol. Patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of a glioblastoma is made. a) Central pathology review is required for study entry. Either H & E stained slides from diagnosis or more recent tumor sampling OR unstained tumor sections must be submitted and reviewed by the study neuropathologist. b) A paraffin-embedded tumor block (preferred) or 15 unstained tumor section slides are required to be submitted at the time of registration.
2. All patients must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients must have signed an authorization for the release of their protected health information. Patients must be registered in the MD Anderson Cancer Center Office of Multicenter Clinical Research (OMCR) database prior to treatment with study drug.
3. Patients must be >/= 18 years old.
4. Patients must have a Karnofsky performance status of >/= 70
5. At the time of registration: Patients must have recovered from the toxic effects of prior therapy: >/= 28 days from any investigational agent, >/= 28 days from prior cytotoxic therapy (>/= 7 days from prior daily administered [i.e. metronomic] cytotoxic agents) , >/= 14 days from vincristine, >/= 42 days from nitrosoureas, >/= 21 days from procarbazine administration, and >/= 7 days for non-cytotoxic agents, e.g., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
6. Patients must have adequate bone marrow function (ANC >/= 1,000/mm3, platelet count of >/= 100,000/mm3, and hemoglobin >/= 10 gm/dl), adequate liver function (SGOT < 2.5 times ULN and bilirubin < 2 times ULN), and adequate renal function (creatinine < 1.5 times ULN) before starting therapy. These tests must be performed within 14 days prior to treatment start date. Eligibility level for hemoglobin may be reached by transfusion.
7. Patients must have shown unequivocal radiographic evidence for tumor progression by MRI or CT scan. A scan should be performed within 14 days prior to treatment start date and on a steroid dose that has been stable or decreasing for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, i.e., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
8. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply: a). They have recovered from the effects of surgery and are at least four weeks from craniotomy or at least 1 week from stereotactic biopsy. b). Residual disease following resection of recurrent GBM is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done no later than 96 hours in the immediate post-operative period or at least 4 weeks post-operatively, within 14 days prior to treatment start date. If the 96-hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
9. Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 12 weeks from the completion of radiation therapy to study entry unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there is histopathologic confirmation of recurrent tumor.
10. Patients with prior therapy that included interstitial brachytherapy or stereotactic radiosurgery must have confirmation of true progressive disease rather than radiation necrosis based upon either PET or Thallium scanning, MR spectroscopy or surgical/pathological documentation of disease.
11. Women of childbearing potential must have a negative B-HCG pregnancy test documented within 14 days prior to treatment start date.
12. Prothrombin time (PT)/international normalized ratio (INR) within normal limits and partial thromboplastin time (PTT) below upper limit of normal.
13. No evidence of hemorrhage on the baseline MRI or CT scan other than those that are stable grade 1.
14. Patients must be at first or second relapse. Relapse is defined as progression following initial therapy (i.e. radiation+/- chemo if that was used as initial therapy). The intent therefore is that patients have no more than 2 prior therapies (initial and treatment for 1 relapse). If the patient had a surgical resection for relapsed disease and no anti-cancer therapy was instituted for up to 12 weeks, and the patient undergoes another surgical resection, this is considered as 1 relapse. For patients who had prior therapy for a low-grade glioma, the surgical diagnosis of a high-grade glioma will be considered the first relapse.

Exclusion Criteria:

1. Current concomitant chemotherapy, radiation therapy, or immunotherapy other than as specified in the protocol.
2. History of coagulation disorder associated with bleeding or thrombotic events.
3. Any significant concurrent disease, illness, or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow up, or interpretation of study results, including legal incapacity or limited legal capacity.
4. Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids
5. Active infection requiring intravenous antibiotics
6. Requires anticoagulation therapy with vitamin K antagonists, heparin, or thrombin or factor X inhibitors. (Low molecular weight heparin is allowed)
7. Have had a diagnosis of another malignancy, unless the patient has been disease-free for at least 12 months following the completion of curative intent therapy, with the following exceptions: a). Patients with treated non-melanoma skin cancer, in situ carcinoma, or cervical intraepithelial neoplasia, regardless of the disease-free duration, are eligible for this study if definitive treatment for the condition has been completed. b). Patients with organ-confined prostate cancer with no evidence of recurrent or progressive disease based on prostate-specific antigen (PSA) values are also eligible for this study if hormonal therapy has been initiated or a radical prostatectomy has been performed.
8. Inability to comply with study and/or follow-up procedures;
9. Current or planned participation in an experimental therapeutic drug study;
10. Severe hepatic insufficiency (ongoing grade 3 or greater hepatic adverse events) or known active chronic hepatitis
11. Prior treatment with cilengitide, bevacizumab or other VEGF/VEGFR-targeting therapy.
12. Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
13. Any prior history of hypertensive crisis or hypertensive encephalopathy
14. New York Heart Association (NYHA) Grade II or greater congestive heart failure
15. History of myocardial infarction or unstable angina within 6 months prior to study enrollment
16. History of stroke or transient ischemic attack within 6 months prior to study enrollment
17. Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
18. Symptomatic peripheral vascular disease
19. Evidence of bleeding diathesis or coagulopathy
20. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
21. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
22. History of abdominal fistula, gastrointestinal perforation, intra-abdominal abscess or endoscopically-proven ulcer (esophageal, gastric or duodenal) within 6 months prior to study enrollment
23. Serious, non-healing wound, ulcer, or bone fracture
24. Proteinuria at screening as demonstrated by either: a). Urine protein:creatinine (UPC) ratio >/= 1.0 at screening OR b). Urine dipstick for proteinuria >/= 2+ (patients discovered to have >/= 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate </= 1g of protein in 24 hours to be eligible).
25. Known hypersensitivity to any component of bevacizumab, Chinese hamster ovary cell products or other recombinant human or humanized antibodies.
26. Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential
27. Known hypersensitivity to cilengitide, other trial treatment(s) or diluents (when applicable), including placebo or other comparator drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | 6 months
  Primary goal is to assess efficacy of administering cilengitide with bevacizumab for treatment of patients with recurrent gliomas who are bevacizumab-naïve. Study is designed to have adequate power to compare the efficacy of the experimental regimen to a historical benchmark. Basis for assessment is proportion of patients who have survived 6 months without disease progression (PFS-6).

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, MD,BS, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org